CLINICAL TRIAL: NCT02674607
Title: the Potential Immunomodulatory Effects of Spirulina on Thalassemic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Professor Mohamed Elshanshory, head of pediatric hematology and oncology unit, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2132/10/13
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients (Experimental): thirty children with beta thalassemia major will receive oral spirulina (tablets=500 mg) for 3 months with a dose of 250 mg/kg/day (maximum dose 4 gm)
  Interventions: Dietary Supplement: Spirulina
- controls (No Intervention): thirty healthy children of matched age and sex

INTERVENTIONS:
Dietary Supplement: Spirulina
  Arms: patients

SUMMARY:
The aim of this study is to evaluate the possible immunologic effects of spirulina in children with beta thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* children with thalassemia major

Exclusion Criteria:

* children with other chronic hemolytic anemias

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
cluster of differentiation (CD4/CD25) ratio | 3 months
cluster of differentiation (CD33/CD11b/Lin) ratio | 3 months
serum immunoglobulins levels | 3 months
serum levels of interferon gamma | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El-Shanshory, MD, Principal Investigator — professor of pediatrics- head of hematooncology unit of pediatric department- Tanta University
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt